CLINICAL TRIAL: NCT02718599
Title: Effect of Terlipressin Infusion on Systemic and Hepatic Hemodynamics During Hepatobiliary Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Magdy Mohammed Mahdy Sayed, Effect of terlipressin and hepatic hemodynamics during hepatobiliary surgery infusion on systemic., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABC-123-DE
Record Dates: First submitted 2016-03-19; First posted 2016-03-24 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2016-03

CONDITIONS: Hemodynamics, Liver, Terlipressin
MeSH Terms: interventions — Terlipressin; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Terlipressin (Active Comparator): Terlipressin will be started at the beginning of surgery as an initial bolus dose of 1 mg over 30 mints(1 mg/50 ml normal saline at a rate of 100 ml/h) followed by a continuous infusion of 2 μg/kg/h(1 mg/50 ml at a rate equal to wt/10 ml per hour) and weaned in the postoperative period over 4 hours.
  Interventions: Drug: terlipressin
- CONTROL (Placebo Comparator): Patients receive the same volume of 0.9% saline in place of terlipressin for the same duration(50 ml normal saline at a rate of 100 ml/h followed by a continuous infusion of 50 ml at a rate equal to wt/10 ml per hour and weaned in the postoperative period over 4 hours).
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: terlipressin — Terlipressin will be started at the beginning of surgery as an initial bolus dose of 1 mg over 30 mints(1 mg/50 ml normal saline at a rate of 100 ml/h) followed by a continuous infusion of 2 μg/kg/h(1 mg/50 ml at a rate equal to wt/10 ml per hour) and weaned in the postoperative period over 4 hours.
  Other Names: glypressin
  Arms: Terlipressin
Drug: normal saline — Patients receive 50 ml normal saline at a rate of 100 ml/h followed by a continuous infusion of 50 ml at a rate equal to wt/10 ml per hour and weaned in the postoperative period over 4 hours.
  Other Names: 0.9 Nacl
  Arms: CONTROL

SUMMARY:
To evaluate the effect of terlipressin infusion on systemic and hepatic hemodynamics during hepatobiliary surgery

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Any gender.
* ASA (American Society of Anesthesiologists) Classification( Class I-II)
* Patients undergoing major elective hepatobiliary surgery.

Exclusion Criteria:

* Preoperative renal failure (GFR < 50 ml/min).
* Severe liver dysfunction (Child- turcotte -Pugh grade C).
* Hyponatremia (<132 mmol/l).
* Severe aortic regurgitation, severe mitral regurgitation, heart failure.
* Symptomatic coronary heart disease.
* Bradycardic arrhythmia (heart rate < 60/min).
* Peripheral artery occlusive disease (clinical stadium II-IV).
* Uncontrolled arterial hypertension (Blood pressure >160/100 mmHg despite intensive treatment).
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
portal pressure changes | intraoperative period
  portal pressure changes in mmHg

SECONDARY OUTCOMES:
Effect on systemic vascular resistance | intraoperative period
  •Effect on systemic vascular resistance in dyne.s/cm5
Renal impairment | for 3 days in the postoperative period
  Number of patients with renal impairment [defined as at least a doubling of serum creatinine or oliguria (<500 mL/24 hours)].
Blood units transfused | intraoperative period
  Number of packed RBCs (red blood cells) units transfused

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Samy, Study Director — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mahdy MM, Abbas MS, Kamel EZ, Mostafa MF, Herdan R, Hassan SA, Hassan R, Taha AM, Ibraheem TM, Fadel BA, Geddawy M, Sayed JA, Ibraheim OA. Effects of terlipressin infusion during hepatobiliary surgery on systemic and splanchnic haemodynamics, renal function and blood loss: a double-blind, randomized clinical trial. BMC Anesthesiol. 2019 Jun 15;19(1):106. doi: 10.1186/s12871-019-0779-6. PMID 31200638